CLINICAL TRIAL: NCT00709995
Title: Dose Finding and Randomized, Multicenter, Placebo-Controlled, Phase 2 Study of Enzastaurin and Sunitinib Versus Placebo and Sunitinib in Patients With Metastatic Renal Cell Carcinoma
Brief Title: A Study for Participants With Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11531; H6Q-MC-S061 (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-06-30; First posted 2008-07-03 (Estimated); Results first posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-01

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — enzastaurin; Sunitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 Arm A: Enzastaurin + Sunitinib (Experimental): (Cohort 1): On cycle 1, day 1 a loading dose 125 milligram (mg) of Enzastaurin was administered by mouth orally, (BID) twice a day, followed by Enzastaurin 125 mg administered, twice a day, Days 2 through 42 of a 6-week cycle.
  (Cohort 2): Cycle 1, Day 1 loading dose 375 mg of Enzastaurin administered po three times a day (TID), followed by 250 mg, po, BID continuously until disease progression, unacceptable toxicity, death, or discontinuation from the study for any other reason.
  Sunitinib 50 mg was administered orally, once daily, Days 1-28, then rest (no drug given) days 29-42.
  Phase 2 (Part 2): Randomized Double-Blind: Dosing was determined by Part 1. Part 2 was not activated per recommendation of safety review committee.
  Enzastaurin: Cycle 1, Day 1 loading dose 375 mg administered orally, (TID) three times a day, followed by Part 1 dose twice a day on Days 2-42 of 6 week cycle.
  Sunitinib: 50 mg administered orally, once daily, on Days 1-28, then rest Days 29-42.
  Interventions: Drug: Enzastaurin; Drug: Sunitinib
- Part 2 Arm B: Sunitinib + Placebo (Placebo Comparator): Part 2 was not activated per recommendation of safety review committee.
  Sunitinib: 50 mg administered orally, once daily, Day 1-28, then rest Days 29-42.
  Placebo: Cycle 1 Day 1 loading dose 3 tablets on Day 1, then 2 tablets daily, days 2-42.
  Interventions: Drug: Sunitinib; Drug: Placebo

INTERVENTIONS:
Drug: Enzastaurin — Administered orally
  Other Names: LY317615
  Arms: Part 1 Arm A: Enzastaurin + Sunitinib
Drug: Sunitinib — Administered orally
Drug: Placebo — Administered orally
  Arms: Part 2 Arm B: Sunitinib + Placebo

SUMMARY:
This study will compare the effects of Enzastaurin plus Sunitinib versus Sunitinib alone in metastatic Renal Cell Cancer.

DETAILED DESCRIPTION:
This is a multicenter, Phase 2 study of enzastaurin and sunitinib versus placebo and sunitinib as first-line therapy in participants with metastatic renal cell carcinoma, containing 2 parts. Part 1 is a safety lead-in study with 12 participants and possible dose escalation. Part 2 is a randomized, double-blind, Phase 2 study in 110 participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants with metastatic Renal Cell Carcinoma (RCC) who have not received prior treatment with systemic (adjuvant or neoadjuvant) therapy for RCC (including targeted therapy such as tyrosine kinase inhibitors or bevacizumab, immunotherapy, chemotherapy, hormonal, or investigational therapy)
* Histologically confirmed RCC with metastases with a component of clear (conventional) cell histology
* Evidence of unidimensional measurable disease, measured by computed tomography (CT) scan or magnetic resonance imaging (MRI)
* Primary tumor has been surgically removed by nephrectomy or nephron-sparing surgery
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Participants must sign an informed consent document

Exclusion Criteria:

* Have received prior treatment with sunitinib or enzastaurin
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* Have had any of the following within 12 months prior to study drug administration:

  * myocardial infarction,
  * severe/unstable angina,
  * coronary/peripheral artery bypass graft,
  * symptomatic congestive heart failure (CHF),
  * cerebrovascular accident,
  * transient ischemic attack, or
  * pulmonary embolism
* Note: Ongoing treatment with therapeutic doses of Coumadin® (warfarin) or a derivative of Coumadin or phenprocoumon is not allowed, but prophylactic, low-dose Coumadin (≤ 2 mg daily) for deep vein thrombosis is allowed. In such cases, prothrombin time/international normalization ratio (PT/INR) should be very closely monitored as clinically indicated
* Ongoing cardiac arrhythmias >New York Health Association Class II, atrial fibrillation of any grade, or prolongation of the QTc interval to >450 millisecond (msec) for males or >470 msec for females.
* Have uncontrolled hypertension [>150/100 millimeter of mercury (mm/Hg) despite optimal medical therapy], or history of poor compliance with antihypertensive treatment
* Require concomitant use of potent Cytochrome P450 3A4 (CYP3A4) inducer, for example, rifampicin or potent CYP3A inhibitors, such as ketoconazole.
* Significant surgery or radiation therapy <4 weeks of starting study treatment. Prior palliative radiotherapy to metastatic lesion(s) is/are permitted, provided there is at least 1 measurable lesion that has not been irradiated
* Participants who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-06-30 (Actual); Primary Completion 2010-02-15 (Actual); Study Completion 2018-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) Mon - Fri 9AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna, Austria
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Villejuif, France
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome, Italy
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part 1 completers finished 3 or more cycles and included those with progressive disease. Part 2 was not performed and was not activated due to sponsor broad decision to not pursue enzastaurin in solid tumors.
Groups:
- Modified Regimen A (Cohort 1): On cycle 1, day 1 a loading dose 125 milligram (mg) of Enzastaurin was administered by mouth orally, (BID) twice a day, followed by Enzastaurin 125 mg administered, twice a day, Days 2 through 42 of a 6-week cycle.
  Sunitinib 50 mg was administered orally, (QD) once daily, Days 1-28, then rest (no drug given) Days 29-42.
- Regimen A (Cohort 2): Enzastaurin was given on Day 1 of Cycle 1 as a loading dose of 1125 mg (3 tablets of 125 mg each, taken 3 times a day with at least 4 hours between doses), followed by daily total dose of 500 mg (2 tablets of 125 mg each, BID) continuously until disease progression, unacceptable toxicity, death, or discontinuation from the study for any other reason.
  Sunitinib 50 mg was administered orally, once daily, Days 1-28, then rest (no drug given) Days 29-42.
Period: Overall Study
Arm/Group | Modified Regimen A (Cohort 1) | Regimen A (Cohort 2)
Started | 11 | 6
Progressive Disease | 6 | 1
Completed | 6 | 1
Not Completed | 5 | 5
Not completed — Adverse Event | 4 | 2
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug in Part 1.
Groups:
- Modified Regimen A (Cohort 1): On cycle 1, day 1 a loading dose 125 milligram (mg) of Enzastaurin was administered by mouth orally, (BID) twice a day, followed by Enzastaurin 125 mg administered, twice a day, Days 2 through 42 of a 6-week cycle Sunitinib 50 mg was administered orally, once daily, Days 1-28, then rest (no drug given) Days 29-42.
- Total: Total of all reporting groups
Arm/Group | Modified Regimen A (Cohort 1) | Regimen A (Cohort 2) | Total
Number analyzed (Participants) | 11 | 6 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (5.44) | 58.5 (8.42) | 59.6 (6.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 6 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 6 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 1 | 1 | 2
  Poland | 6 | 4 | 10
  Italy | 3 | 0 | 3
  France | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) in Part 2
Description: Progression-free survival (PFS) was defined as the number of months between the date of randomization and the date of first documented disease progression or the date of death due to any cause, whichever came first.
Time Frame: Randomization to Measured Progressive Disease (PD) (Up to 24 Months)
Population: Zero participants data were collected. Part 2 was not activated due to sponsor broad decision to not pursue Enzastaurin in solid tumors.
Groups:
- Enzastaurin + Sunitinib: Enzastaurin: Cycle 1, Day 1 loading dose 375 mg administered orally, (TID) three times a day, followed by Part 1 dose twice a day on Days 2-42 of 6-week cycle.
  Sunitinib: 50 mg administered orally, once daily, on Days 1-28, then rest Days 29-42.
- Sunitinib + Placebo: Sunitinib: 50 mg administered orally, once daily, Day 1-28, then rest Days 29-42.
  Placebo: Cycle 1 Day 1 loading dose 3 tablets on Day 1, then 2 tablets daily, Days 2-42.
Arm/Group | Enzastaurin + Sunitinib | Sunitinib + Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Survival (OS) in Part 2
Description: OS time was defined as the number of months between the date of randomization and the date of death due to any cause.
Time Frame: Randomization to Death from Any Cause (Up to 24 Months)
Population: Zero participant data were collected. Part 2 was not activated due to sponsor broad decision to not pursue Enzastaurin in solid tumors.
Groups:
- Enzastaurin + Sunitinib: Enzastaurin: Cycle 1, Day 1 loading dose 375 mg administered orally, three times a day, followed by Part 1 dose twice a day on Days 2-42 of 6-week cycle.
  Sunitinib: 50 mg administered orally, once daily, on Days 1-28, then rest Days 29-42.
Arm/Group | Enzastaurin + Sunitinib | Sunitinib + Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time-To-Tumor Progression in Part 2
Description: Time to tumor progression (TTP) at initial treatment was defined as the number of months between date of randomization and the date of first documented disease progression or the date of death due to disease under study, whichever came first.
Time Frame: Randomization to the Date of Objective Progressive Disease or Date of Death due to Study Disease, whichever came first (Up to 24 Months)
Population: as for outcome 2
Arm/Group | Enzastaurin + Sunitinib | Sunitinib + Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Adverse Events (AEs) or Serious AEs (SAEs) in Part 1
Description: Clinically significant events were defined as serious adverse events, regardless of causality. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Event module.
Time Frame: Randomization to Study Completion (Up to 6 Cycles)
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Modified Regimen A (Cohort 1) | Regimen A (Cohort 2)
Number analyzed (Participants) | 11 | 6
Participants
  AEs | 11 | 6
  SAEs | 3 | 1

5. Secondary Outcome: Pharmacokinetics (PK): Area Under Concentration Time Curve During One Dosing Interval at Steady State (AUCτ,ss) of Enzastaurin + Metabolite (LSN326020) + Total Analytes in Part 1
Description: Pharmacokinetics (PK) was assessed in participants to determine the area under the concentration time curve during one dosing interval at steady state (AUCτ,ss) of Enzastaurin, LSN326020 and total Analytes. τ equals 12 hours for Enzastaurin, LSN326020 and total Analytes.
Time Frame: Cycle 1 Day 15: Predose, 2, 4, and 6 - 8 hours, Up to 12 Hours Post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole*hour/liter (nmol*hr/L)
Arm/Group | Modified Regimen A (Cohort 1) | Regimen A (Cohort 2)
Number analyzed (Participants) | 11 | 5
nanomole*hour/liter (nmol*hr/L)
  Enzastaurin | 12000 (144) | 22600 (91)
  LSN326020 | 8820 (76) | 12200 (73)
  Total Analytes | 21400 (101) | 35200 (82)

6. Secondary Outcome: PK: Maximum Concentration at Steady State (Cmax,ss) of Enzastaurin + LSN326020 + Total Analytes in Part 1
Description: PK was assessed in participants to determine the maximum concentration at steady state (Cmax, ss) of Enzastaurin + LSN326020 + total analytes.
Time Frame: Cycle 1 Day 15: Predose, 2, 4, and 6 - 8 hours, Up to 12 Hours Post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole/liter (nmol/L)
Arm/Group | Modified Regimen A (Cohort 1) | Regimen A (Cohort 2)
Number analyzed (Participants) | 11 | 5
nanomole/liter (nmol/L)
  Enzastaurin | 1310 (109) | 2650 (71)
  LSN326020 | 816 (72) | 1140 (64)
  Total Analytes | 2130 (88) | 3740 (65)

ADVERSE EVENTS:
Time Frame: From Baseline to Study Completion (Up to 123 Months)
Description: All participants who received at least one dose of study drug in Part 1.
Groups:
- Modified Regimen A (Cohort 1): On cycle 1, day 1 a loading dose 125 milligram (mg) of Enzastaurin was administered by mouth orally, (BID) twice a day, followed by Enzastaurin 125 mg administered, twice a day, Days 2 through 42 of a 6-week cycle.
  Sunitinib 50 mg was administered orally, once daily, Days 1-28, then rest (no drug given) Days 29-42.
- Regimen A (Cohort 2): Enzastaurin was given on Day 1 of Cycle 1 as a loading dose of 1125 mg (3 tablets of 125 mg each, taken 3 times a day with at least 4 hours between doses), followed by daily total dose of 500 mg (2 tablets of 125 mg each, BID) continuously until disease progression, unacceptable toxicity, death, or discontinuation from the study for any other reason
  Sunitinib 50 mg was administered orally, once daily, Days 1-28, then rest (no drug given) Days 29-42.
Arm/Group | Modified Regimen A (Cohort 1) | Regimen A (Cohort 2)
Serious Adverse Events (participants affected / at risk) | 3/11 | 1/6
Other Adverse Events (participants affected / at risk) | 11/11 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modified Regimen A (Cohort 1) (N=11) | Regimen A (Cohort 2) (N=6)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Modified Regimen A (Cohort 1) (N=11) | Regimen A (Cohort 2) (N=6)
Anaemia (Blood and lymphatic system disorders) | 8 (33) | 4 (10)
Leukopenia (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 5 (7) | 1 (87)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (20) | 2 (32)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (3) | 1 (1)
Eyelid oedema (Eye disorders) | 2 (2) | 0 (0)
Lacrimation increased (Eye disorders) | 2 (5) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal inflammation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dental discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (14) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (7) | 2 (3)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 6 (9) | 1 (4)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (8)
Asthenia (General disorders) | 3 (5) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (2) | 0 (0)
Face oedema (General disorders) | 1 (1) | 1 (5)
Fatigue (General disorders) | 5 (5) | 3 (9)
General physical health deterioration (General disorders) | 2 (2) | 1 (2)
Influenza like illness (General disorders) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 4 (7) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (13)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (60)
Blood amylase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin decreased (Investigations) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 3 (22)
Blood lactate dehydrogenase increased (Investigations) | 1 (2) | 0 (0)
Blood sodium increased (Investigations) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (31)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 1 (2) | 0 (0)
Vitamin b12 decreased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 4 (4) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (7) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Dysgeusia (Nervous system disorders) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (5) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 5 (7) | 2 (3)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria localised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Yellow skin (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Part 1 completers finished 3 or more cycles and included those with progressive disease. Part 2 was not performed and was not activated due to sponsor broad decision to not pursue enzastaurin in solid tumors

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days